CLINICAL TRIAL: NCT01181635
Title: Can Psychotherapy Reduce Sickness Absence?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lovisenberg Diakonale Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010/494 (REK)
Record Dates: First submitted 2010-08-12; First posted 2010-08-13 (Estimated); Last update posted 2019-08-09 (Actual); Status verified 2016-04

CONDITIONS: Mental Disorders
MeSH Terms: conditions — Mental Disorders | interventions — Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Psychotherapy (Experimental): Short-term pychotherapy and/or psychoeduchative courses.
  Interventions: Behavioral: Psychotherapy

INTERVENTIONS:
Behavioral: Psychotherapy — Standard psychotherapy for psychiatric disorders.

SUMMARY:
The purpose of this study is to examine if psychotherapy can reduce sickness absence.

DETAILED DESCRIPTION:
Sickness absence due to psychiatric problems is considered a growing problem in Norway. Little research is done to examine if psychotherapy can reduce sickness absence. Since 2007 there is a government sponsored program in Norway (Raskere tilbake) aimed at reducing sickness absence. This study examines if psychotherapy within this program, delivered at an out-patient clinic, actually reduces sickness absence. Levels of absenteeism is measured before, after and 6 months after treatment. This is a quasi-experimental study, where the treatment-group will be compared with a statistical group in the general population, that is socio-demographical similar and has similar history of sickness absence but haven't been to treatment. Changes in levels of symptoms and quality of life will also be measured. The participants will be asked to describe their working environment, and this will be related to outcome-measures.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving psychotherapy at Lovisenberg DPS/Raskere Tilbake

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2010-08; Primary Completion 2019-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Sickness absence | Before, after and 6 months after treatment.
  Present status (working or sick).

SECONDARY OUTCOMES:
Psychiatric symptoms | Before, after and 6 months after treatment.
  CORE-OM.
Quality of life (QALY) | Before, after and 6 months after treatment.
  15 D

CONTACTS AND LOCATIONS:
Overall Officials: Bjørn Lau, phd, Study Director — Lovisenberg Diakonale Hospital
Locations (1):
- Lovisenberg diakonale sykehus, Lovisenberg DPS, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Victor M, Lau B, Ruud T. Predictors of Return to Work 6 Months After the End of Treatment in Patients with Common Mental Disorders: A Cohort Study. J Occup Rehabil. 2018 Sep;28(3):548-558. doi: 10.1007/s10926-017-9747-5. PMID 29234955
- [Derived] Victor M, Lau B, Ruud T. Predictors of return to work among patients in treatment for common mental disorders: a pre-post study. BMC Public Health. 2017 Jul 18;18(1):27. doi: 10.1186/s12889-017-4581-4. PMID 28720129